CLINICAL TRIAL: NCT03200496
Title: Comparisons of Pharmacokinetics and Safety/Tolerability Profiles Between DA-5206 and Talion® Under Fasting and Fed States in Healthy Male Subjects
Brief Title: Pharmacokinetics and Safety/Tolerability Profiles of DA-5206 Versus Talion® Under Fasting and Fed States in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA5206_BE_Ⅰ
Record Dates: First submitted 2017-06-26; First posted 2017-06-27 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TALION® (Experimental)
  Interventions: Drug: TALION®
- DA-5206(Fasting) (Experimental)
  Interventions: Drug: DA-5206(Fasting)
- DA-5206(Fed) (Experimental)
  Interventions: Drug: DA-5206(Fed)

INTERVENTIONS:
Drug: DA-5206(Fasting) — Test drug l : DA-5206(Fasting)
  Arms: DA-5206(Fasting)
Drug: DA-5206(Fed) — Test drug ll : DA-5206(Fed)
  Arms: DA-5206(Fed)
Drug: TALION® — Reference drug : Talion®
  Arms: TALION®

SUMMARY:
This is Open-label, Randomized, 3-sequence study to compare of pharmacokinetics and safety/tolerability profiles betweens DA-5206, a SR formulation of bepotastine besilate and Talion®, a IR formulation of bepotastine besilate under fasting and fed states in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer 19 years to 45 years
* Body mass index in the range of 18 to 29 kg/m2 and body weight greater than 50 kg
* The subjects personally signed and dated informed consent document after informed of all pertinent aspects of the study, fully understanding and determided spontaneously to participate

Exclusion Criteria:

* Subject with serious active cardiovascular, respiratory, hepatologic, renal, hematologic, endocrine, urologic, immunologic, dermal, neurologic, or psychological disease or history of such disease
* Subject with acute disease within 28 days before the first dose of Investigational product
* Subject with known for history of disease which affect on the absorption, distribution, metabolism, excretion of drug
* Subjects who are unwilling or unable to use highly effective methods of contraception as outlined in this protocol for the duration of the study

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 0~24hr
  PK Parameter
Peak Plasma Concentration (Cmax) | 0~24hr
  PK Parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea